CLINICAL TRIAL: NCT04775225
Title: Hip Denervation in Juvenile Idiopathic Arthritis
Brief Title: Hip Denervation in Juvenile Idiopathic Arthritis With Hip Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3012020
Record Dates: First submitted 2021-02-17; First posted 2021-03-01 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Juvenile Idiopathic Arthritis; Hip Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Lidocaine; Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hip denervation group (Active Comparator): This group will receive Lidocaine 2% block of the femoral and obturator genicular branches.
  Interventions: Drug: Lidocaine
- control group (Placebo Comparator): this group will receive saline injection subcutaneously at the same places.
  Interventions: Drug: Placebo
- Steroid (Active Comparator): This group with receiving an intra-articular injection of 80mg triamcinolone
  Interventions: Drug: Steroid

INTERVENTIONS:
Drug: Lidocaine — denervation of the obturator and femoral genicular branches by Lidocaine 2 %
  Other Names: The active denervation group
  Arms: Hip denervation group
Drug: Placebo — an equivalent amount of saline will be injected subcutaneously in 2 points similar to the active group
  Other Names: The control group
  Arms: control group
Drug: Steroid — Intra-articular injection of 80mg of triamcinolone
  Other Names: The active steroid group
  Arms: Steroid

SUMMARY:
Patients having juvenile idiopathic arthritis (according to ILAR criteria) with hip arthritis were divided into 3 groups. Group 1 received hip denervation and group 2 controlled and received a subcutaneous injection of saline, and group 3 received intra-articular triamcinolone. Outcome measures included pain, tenderness, range of motion, SOLAR, HARISS score. These outcomes were measured at baseline, 2 weeks, and 16 weeks

DETAILED DESCRIPTION:
The aim of the study is to test the effect of denervation of the active hip in JIA and compare it with a placebo without changing systemic treatment during the study. Outcome measures included pain, range of motion, SOLAR score, and Harris functional score.

ELIGIBILITY:
Inclusion Criteria:

* patients with JIA with unilateral hip arthritis

Exclusion Criteria:

* hip involvement due to other causes including
* septic arthritis
* other connective tissue diseases
* Avascular necrosis

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale | Baseline, 2 weeks and 16 weeks
  a scale from 0-100 will be used 0 means no pain 100 means the maximum pain
Change in range of motion | Baseline, 2 weeks and 16 weeks
  flexion, internal rotation, external rotation range will be calculated
Change in Harris functional score | Baseline, 2 weeks and 16 weeks
  100 means best results and 0 means worst results
semiquantitative tenderness score | Baseline, 2 weeks and 16 weeks
  0 means no tenderness and 3 means maximum tenderness
Change in SOLAR score | Baseline, 2 weeks and 16 weeks
  GSUS. 0 means the least synovitis and the maximum, PDUS, o means no PD and 3 the maximum

CONTACTS AND LOCATIONS:
Locations (1):
- ahmed Elsaman, Sohag, Egypt